CLINICAL TRIAL: NCT02949960
Title: DMT210 Topical Gel in the Treatment of Mild to Moderate Atopic Dermatitis
Brief Title: DMT210 Topical Gel in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermata Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMT210-002
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Dermatitis; Skin Diseases; Skin Diseases, Genetic; Dermatitis, Atopic; Skin Diseases, Eczematous; Hypersensitivity; Immune System Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases; Skin Diseases, Genetic; Skin Diseases, Eczematous; Hypersensitivity; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMT210 Topical Gel (Experimental): DMT210 Topical Gel 5% applied to target lesion twice daily
  Interventions: Drug: DMT210 Topical Gel
- Vehicle Control (Placebo Comparator): Topical Gel vehicle applied to target lesion twice daily
  Interventions: Drug: Vehicle Control

INTERVENTIONS:
Drug: DMT210 Topical Gel — DMT210 Topical Aqueous Gel 5% applied twice daily
  Arms: DMT210 Topical Gel
Drug: Vehicle Control — Topical Vehicle Gel applied twice daily
  Arms: Vehicle Control

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of DMT210 Gel, 5% compared to vehicle control following 28 days of twice-daily topical application to selected target lesions in male and female patients with mild to moderate atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 12 years or older
* Patient has chronic, stable AD that has been present for at least 3 months with 5-35% (inclusive) BSA (Body Surface Area) of AD involvement
* Patient has two analogous, Target Lesions; one lesion within each of the two Treatment Areas
* Patient is willing and able to comply with the protocol

Exclusion Criteria:

* Patient has used topical therapies for AD within the Treatment Areas 2 weeks before baseline

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
ADSI (Atopic Dermatitis Severity Index) score of each Target lesion | Day 28
  Change from baseline in ADSI score between Vehicle and 5% gel

SECONDARY OUTCOMES:
Individual Signs and Symptoms of Atopic Dermatitis of each Target Lesion | Day 28
  Change from baseline in AD symptom scores between Vehicle and 5% gel
Investigator Global Assessment (IGA) of the Treatment Area | Day 28

OTHER OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nardo, PhD, Study Director — Dermata Therapeutics
Locations (2):
- United States (2):
  - Dermata Investigational Site, Houston, Texas
  - Dermata Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No